CLINICAL TRIAL: NCT05611502
Title: A Combined Neurofeedback- TMS Intervention for Alcohol Use Disorder - Aim 2
Brief Title: Influence of TMS on Attention Modulation
Acronym: TAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Samantha Fede, Assistant Professor, Auburn University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 21510; R00AA027830 (NIH)
Record Dates: First submitted 2022-10-26; First posted 2022-11-10 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Drinking, Alcohol
Keywords: alcohol; attention; TMS; binge drinking; emotion; social cognition; moral; MRI; frontal eye fields; moral cognition
MeSH Terms: conditions — Alcohol Drinking; Binge Drinking

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive each arm in counterbalanced order (AB or BA).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TMS A (Experimental): TMS administered over right frontal eye field at 10 Hz, 110% of MT, 60 x 5 sec trains, 25 sec ITI
  Interventions: Device: TMS
- TMS B (Active Comparator): TMS administered over right frontal eye field at 1 Hz, 110% of MT, 7 x 225 sec trains, 30 sec ITI
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — TMS will be administered in a pattern that is either excitatory or inhibitory.
  Other Names: Magventure MagPro

SUMMARY:
The purpose of this study is to help understand how attention processes influence brain engagement during emotion and social cognition. The investigators also want to know if these processes are associated with drinking alcohol.

Participation includes three study visits of about 2 hours each over approximately a month. The first visit involves a magnetic resonance imaging (MRI) scan and answering survey questions. Each of the next two visits will involve a session of transcranial magnetic stimulation (TMS, a non-invasive brain stimulation technique) followed by another MRI scan.

People in the Auburn/Opelika area 19 or older are eligible to participate. People who drink alcohol and people who do not drink or don't drink very much are invited to participate.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or Older

2A. (Drinker Group): Reports consuming 4 [if female]/ 5 [if male] or more standard drinks on one occasion at least 2 times a month AND/OR reports consuming more than 7 [if female]/ 14 [if male] standard drinks per week on average

2B. (Healthy Volunteer Group): Reports consuming 4 [if female]/ 5 [if male] or more standard drinks on one occasion less than once a month AND reports consuming less than 7 [if female]/ 14 [if male] standard drinks per week on average

Exclusion Criteria:

1. MRI Contraindications

   1. Presence of metal in the body that would make having a 7T MRI unsafe (including facial tattoos)
   2. Claustrophobia, such that individual would be unable to stay in the MRI for up to 1 hr
   3. Hearing loss, including tinnitus, that might be made worse by MRI or TMS
2. TMS Contraindications

   1. Has ever had a seizure, or has a family history of epilepsy
   2. Taking medications or substances that lower the seizure threshold*
   3. Implanted devices that are in the head or rely on physiological signals
   4. History of neurological disease, such as stroke or brain tumor
   5. Head injury with loss of consciousness greater than 30 minutes
   6. Actively withdrawing from alcohol
3. Family history of schizophrenia or presence of psychotic symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in attention switching | Baseline, immediately following TMS A, immediately following TMS B
  MRI Task- analysis of behavioral data
Change in sociomoral attention switching | Baseline, immediately following TMS A, immediately following TMS B
  MRI Task- analysis of behavioral data
Change in cue reactivity | Baseline, immediately following TMS A, immediately following TMS B
  MRI Task- analysis of behavioral data

SECONDARY OUTCOMES:
Change in brain activity attention switching | Baseline, immediately following TMS A, immediately following TMS B
  MRI Task- analysis of imaging (fMRI) data
Change in brain activity during sociomoral attention switching | Baseline, immediately following TMS A, immediately following TMS B
  MRI Task- analysis of imaging (fMRI) data
Change in brain activity during cue reactivity | Baseline, immediately following TMS A, immediately following TMS B
  MRI Task- analysis of imaging (fMRI) data

CONTACTS AND LOCATIONS:
Overall Officials: Samantha J Fede, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the NIAAA Data Archive according to standard NIAAA procedures. This will include deidentified behavioral, self-report, and imaging data.
  Participants will have the option to opt out of having their individual data available.
Supporting Information: Study Protocol, ICF